CLINICAL TRIAL: NCT00438243
Title: Pilot Study of the Effect of Topical Bromfenac Ophthalmic Solution 0.09%in Patients With Acute Post-operative Cystoid Macular Edema.
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Principal Investigator left institution
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 8377
Record Dates: First submitted 2007-02-21; First posted 2007-02-22 (Estimated); Last update posted 2016-07-04 (Estimated); Status verified 2016-07

CONDITIONS: Cystoid Macular Edema
Keywords: Pseudophakic macular edema
MeSH Terms: conditions — Macular Edema | interventions — bromfenac

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Placebo Comparator): 1 drop affected eye twice daily.
  Interventions: Drug: Refresh Plus
- 2 (Experimental): Bromfenac (Xibrom) 1 drop to affected eye twice a day.
  Interventions: Drug: Bromfenac (Xibrom)

INTERVENTIONS:
Drug: Bromfenac (Xibrom) — 1 drop to affected eye twice daily.
  Arms: 2
Drug: Refresh Plus — 1 drop in the affected eye twice daily
  Arms: 1

SUMMARY:
This research is being done to look at the effects of Bromfenac, also called Xibrom for the treatment of swelling in the retina (the light sensitive tissue in the back of the eye) called "macular edema" that occurs after cataract surgery. Swelling in the retina can lead to blurry vision.

The most commonly used treatment is eyedrops that decrease inflammation and may help stop some of the swelling. The investigators want to see if the drug Bromfenac(Xibrom) can decrease the swelling in the retina after cataract surgery and improve vision in these patients.

DETAILED DESCRIPTION:
Over 2.5 million cataract surgeries are performed yearly in the United States. Despite advances in cataract surgery, cystoid macular edema (CME) is the most common cause of loss of vision after cataract surgery, occurring in approximately 0.3% to 3% of all uncomplicated surgeries. If the surgery is complicated, CME can occur in up to 20% of these patients. In CME, fluid accumulates in cystic spaces within the outer plexiform layer of the retina, resulting in decreased vision.

Ocular nonsteroidal anti-inflammatory drugs (NSAIDs) have been widely used in the treatment of CME. NSAIDs decrease inflammation and are hypothesized to decrease the production of prostaglandins via selective inhibition of the cyclooxygenase pathway, which can result in CME. The standard of care for management of postoperative pseudophakic macular edema to some extent remains unclear. There is currently no FDA-approved therapy for the prophylaxis or treatment of postoperative cystoid macular edema.

Bromfenac (Xibrom)an NSAID and is FDA-approved for ocular use to treat pain and inflammation after ocular surgery. Therefore, these medications might decrease inflammation and be effective in treating CME. The investigators plan to conduct a controlled study to investigate the effect of Bromfenac (Xibrom)in patients who develop CME after cataract surgery. The results of this study may be important in better understanding the pathogenesis and treatment of acute postoperative cystoid macular edema to prevent chronic vision loss.

ELIGIBILITY:
Inclusion Criteria:

* Adults (ages 18 years or older)
* Best-corrected visual acuity 20/40 or worse
* Pseudophakic CME in the study eye with onset at least three weeks and no more than four months after cataract surgery, as document on fluorescein angiography and/or OCT (central subfield >/= 250 microns)
* Agree to avoid disallowed medications (including ocular, topical, or systemic NSAIDs; ocular, topical, or systemic corticosteroids; ocular prostaglandin analogs) throughout the duration of the study. Agree to a 14 day washout period prior to enrollment if currently using a disallowed medication.

Exclusion Criteria:

* History of a known hypersensitivity to bromfenac, or any component of the test agents and/or "procedural" medications (such as anesthetic, dilating drops, fluorescein, etc)
* History of pre-existing macular disease that confounds and/or precludes the evaluation of cystoid macular edema (including but not limited to macular hole, epiretinal membrane with pseudohole, diabetic macular edema, neovascular age-related macular degeneration, acute posterior uveitis)
* CME due to other etiologies such as vein occlusion
* Use of a topical ophthalmic prostaglandin analog within 14 days prior to enrollment, i.e., the subject does not agree to a 14 day washout period prior to enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-05; Primary Completion 2010-07 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects improving >/= 10 letter (2 lines) of best-corrected distance visual acuity at day 90 ± 14 days after initiation of one of the test agents. | 6 months

SECONDARY OUTCOMES:
Analysis of the decrease in the center point retinal thickness by Optical Coherence Tomography (OCT) at 90 ± 14 days after initiation of the test agent. | 6 months
Analysis of patient comfort during the use of test agent as assessed with the ocular comfort grading scale | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Alisa Kim, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- The Johns Hopkins Hospital, Baltimore, Maryland, United States